CLINICAL TRIAL: NCT05090709
Title: Analysis of a Spinal Mobilisation Intervention in People With Multiple Sclerosis
Brief Title: MS Spinal Mobilisation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edinburgh Napier University (Other)
Collaborators: Scottish Hospital Endowments Research Trust (Other); Pacla Medical Limited (Industry)
Responsible Party: Principal Investigator, Rebecca Hamilton, Principal Investigator, Edinburgh Napier University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MS_2
Record Dates: First submitted 2021-09-05; First posted 2021-10-25 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; myometer; muscle stiffness; spinal mobilisations; body sway; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: Mixed factor: between-subject, repeated measures (mobilisation intervention vs general massage).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental A - Mobilisation Intervention (Experimental): Participants receive 4 separate treatment sessions of the 30 minute spinal mobilisation intervention.
  Interventions: Other: Spinal Mobilisation Intervention
- Experimental B - General Massage (Active Comparator): Participants receive 4 separate treatment sessions of the 30 minute general massage.
  Interventions: Other: General Massage

INTERVENTIONS:
Other: Spinal Mobilisation Intervention — 30 minutes spinal mobilisations, rate = 0.37Hz, 22 beats per minute, force = less than grade 1, threshold of 80N, location = L1-L5.
  Arms: Experimental A - Mobilisation Intervention
Other: General Massage — 30 minutes manual touch with no specifications or recordings on rate, pressure or location of touch.
  Arms: Experimental B - General Massage

SUMMARY:
The objective of the study is to measure the effect of a spinal mobilisation intervention on para-spinal muscle tissue quality, functional balance measures, pain and fatigue in people with multiple sclerosis. The mobilisation intervention group will be compared to a general massage group to analyse the difference between the specificities of the intervention compared to general manual touch. Participants will be randomly allocated to a group condition for a between-subject, repeated measures study. The study hypothesises a decrease in lumbar stiffness, body sway, pain and fatigue post the intervention compared to the general massage group.

DETAILED DESCRIPTION:
The long term management of multiple sclerosis (MS) symptoms may often involve manual therapeutics due to observed improvements in muscle stiffness, pain, fatigue and balance. Though these improvements are often anecdotal without objective measurement and without analysis of the manual therapeutic. This is partly due to the vast array of manual therapeutics available as well as the many possible influencing factors contributing to these symptoms.

The objective of this study is to measure and analyse the cumulative effect of a spinal mobilisation intervention on muscle tissue quality, functional balance, pain and fatigue in people with MS. The intervention will be analysed at a specific rate, pressure and location and compared to a general manual touch session with no specificities on rate, pressure or location. Both therapy sessions will be 30 minutes long. The force of both therapy sessions will be recorded in real time by monitoring the vertical ground reaction force (GRF) profile using 2 Kistler force plates placed underneath the treatment plinth. A 0 force will be generated once each participant is lying supine and still on the plinth and recordings will be taken in 30 second samples during the treatment sessions. The summation of the vertical GRFs will be graphed and monitored to check consistency of the treatment force. The mobilisation intervention will be given at a rate of 0.37Hz (22 beats per minute) maintained by a metronome on silent within view of the therapist, the pressure will be maintained at a pressure grade of less than 1 (equal to a threshold of 80N), and maintained consistent physical contact on paraspinal region within L1-L5. The general massage will be applied on the mid-lower back, with no specificities or consistencies; physical contact, rate and force magnitude will not be kept constant. This will be tested on 20 participants with MS who are randomly allocated to a group condition for a between-subject, repeated measures study.

Participants will be randomly allocated to either an intervention or general massage group for which they will attend 4 separate therapy sessions. During the 1st session, the participants will carry out tests for lumbar muscle response, measured stiffness, tone and elasticity (using MyotonPro), functional balance measures in a single-leg balance and sit-to-stand tests (using Kistler force plates), self-reported pain and self-reported fatigue for pre and post treatment sessions. During the subsequent 3 sessions, the participants will complete tests for the myometer, balance and pain post the treatment sessions, and the final fatigue test will be completed after their last session. Participants will therefore complete 5 set of tests for the myometer, balance and pain and the fatigue test is completed pre and post all therapy sessions due to the set-up of the questionnaire.

Participants will complete an online questionnaire before their 1st to screen for eligibility criteria and collect anthropometric details and information on their MS condition. This will be analysed with the results into descriptive statistics and summarised into mean, range and dispersion values. All dependent variables measured for muscle tissue response, functional balance, pain and fatigue will be analysed in between-subject repeated measured ANOVA to determine differences between the 2 treatment groups and between the different treatment time points. Pearson correlations will be carried out on the myometer variables to compare the baseline values to the level of change after their final session due to previously found significant correlations.

More participants were intended for recruitment in the study, a post-hoc power calculation revealed a power of 0.9 with an alpha level at 0.05 with a range of large effect sizes in the results.

ELIGIBILITY:
Inclusion Criteria:

* Must have Multiple Sclerosis diagnosis.
* Must be able to walk independently.
* Must have an EDSS score of 6 or below.

Exclusion Criteria:

Respond positively to any absolute contraindications for spinal manual therapy including:

* segment instability
* infectious disease
* osteomyelitis
* bone tumours
* severe haemophilia
* spinal cord damage
* cervical arterial dysfunction

Respond positively to any relative contraindications for spinal manual therapy including:

* spinal disc prolapse
* spondylosis
* inflammatory arthritides
* osteoporosis
* hypermobile syndrome
* pregnancy
* pregnancy
* cancer
* cardiovascular disease
* respiratory disease
* healing injury
* adverse reaction to previous spinal treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Edinburgh Napier University, Edinburgh, County, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data sets that underlie the results for publication will be shared on a raw data set. This includes the anthropometric data, MS information data, myometer data, functional balance data, pain and fatigue data.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be entered when the study is completed and remain until 1 year post publication of summary data.
Access Criteria: the anonymised participant data underlying the summary data published will be shared on the Edinburgh Napier University University Repository with submission of PhD thesis.
URL: http://researchrepository.napier.ac.uk/Output/2709099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.69) | 39.4 (8.33) | 42.1 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height (m) [Mean (Standard Deviation); unit: meters] | 1.71 (0.09) | 1.72 (0.1) | 1.72 (0.09)
Mass (kg) [Mean (Standard Deviation); unit: Kilograms] | 80.01 (29.89) | 81.15 (26.57) | 80.58 (27.53)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms/meters^2] | 26.95 (8.48) | 26.95 (7.29) | 26.95 (7.61)
Expanded Disability Status Scale [Mean (Standard Deviation); unit: Units on a scale] — Self-reported by participant using pre-screening online survey based on disabilities associated with multiple sclerosis. Scale ranges from 0-10 in 0.5 increments each representing a higher level of disability. 0 represents no disability, 1-4.5 represents people who are able to walk without an aid, 5-9.5 represents more severly disabled and impairment to walking and 10 represents death due to multiple sclerosis complications.
  Units on a scale | 2.45 (0.86) | 2.15 (0.75) | 2.3 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Participant Muscle Stiffness Measure
Description: Myometer measured stiffness taken from Erector Spinae muscle central belly via accelerometer probe registering response from a series of low force mechanical impulses applied perpendicular to the muscle. The muscle central belly was palpated while asking the participant to lift their head and feet at the same time while lying in prone position contracting this muscle. Measurements taken from a myometer device given in Newton-metre units. Further method details are given in the Protocol Document in attachments.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Newton-metres
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Newton-metres | 350.83 (51.54) | 240.07 (18.51)

2. Primary Outcome: Participant Muscle Stiffness Measure
Description: as for outcome 1
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Newton-metres
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Newton-metres | 306.27 (27.41) | 234.77 (22.08)

3. Primary Outcome: Participant Muscle Stiffness Measure
Description: as for outcome 1
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Newton-metres
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Newton-metres | 306.47 (39.87) | 232.37 (24.08)

4. Primary Outcome: Participant Muscle Stiffness Measure
Description: as for outcome 1
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Newton-metres
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Newton-metres | 340.87 (51.27) | 235.33 (27.54)

5. Primary Outcome: Participant Muscle Stiffness Measure
Description: as for outcome 1
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Newton-metres
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Newton-metres | 324.37 (46.21) | 220.27 (17.4)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Stiffness values were analysed as a percentage change from baseline measurements to normalise group variances; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Stiffness values were analysed as a percentage change from baseline measurements to normalise group variances; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

6. Primary Outcome: Participant Single Leg Stance Body Sway Path Length
Description: Force plate recording from single leg stance balance test automatically outputted by software using centre of pressure recording to track position total body sway travelled. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 495.22 (57.12) | 619.57 (77.36)

7. Primary Outcome: Participant Single Leg Stance Body Sway Path Length
Description: as for outcome 6
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 458.45 (51.23) | 524.29 (65.21)

8. Primary Outcome: Participant Single Leg Stance Body Sway Path Length
Description: as for outcome 6
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 387.23 (52.1) | 543.4 (73.15)

9. Primary Outcome: Participant Single Leg Stance Body Sway Path Length
Description: as for outcome 6
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 386.32 (40.55) | 509.36 (51.12)

10. Primary Outcome: Participant Single Leg Stance Body Sway Path Length
Description: as for outcome 6
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 389.22 (55.6) | 491.92 (58.75)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis

11. Primary Outcome: Participant Sit-to-Stand Velocity
Description: Force plate recording from sit-to-stand test.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 160.66 (11.95) | 156.41 (20.78)

12. Primary Outcome: Participant Sit-to-Stand Velocity
Description: Force plate recording from sit-to-stand test.
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 176.01 (12.95) | 142.65 (14.04)

13. Primary Outcome: Participant Sit-to-Stand Velocity
Description: Force plate recording from sit-to-stand test.
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 189.25 (13.77) | 158.36 (14.61)

14. Primary Outcome: Participant Sit-to-Stand Velocity
Description: Force plate recording from sit-to-stand test.
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 166.07 (19) | 131 (9.38)

15. Primary Outcome: Participant Sit-to-Stand Velocity
Description: Force plate recording from sit-to-stand test.
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 164.18 (18.13) | 145.06 (13.76)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Sit-to-stand velocity values were analysed as a percentage change from baseline measurements to normalise group variances; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

16. Primary Outcome: Participant Pain Score - Visual Analogue Scale (VAS)
Description: Self-reported pain score annotated by participant pointing on the VAS sheet. Score is between 0-10 with 0 as lowest pain score and 10 as highest pain score.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 1.2 (0.57) | 0.8 (0.59)

17. Primary Outcome: Participant Pain Score - Visual Analogue Scale (VAS)
Description: as for outcome 16
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 0.5 (0.31) | 0.7 (0.6)

18. Primary Outcome: Participant Pain Score - Visual Analogue Scale (VAS)
Description: as for outcome 16
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 0.6 (0.34) | 0.4 (0.22)

19. Primary Outcome: Participant Pain Score - Visual Analogue Scale (VAS)
Description: as for outcome 16
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 0.6 (0.34) | 0.67 (0.21)

20. Primary Outcome: Participant Pain Score - Visual Analogue Scale (VAS)
Description: as for outcome 16
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 0.5 (0.31) | 0.3 (0.21)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

21. Primary Outcome: Participant Fatigue Score - 5 Item Modified Fatigue Impact Scale.
Description: Self-reported fatigue score from filling out 5 questions on the fatigue questionnaire with possible answers ranging from 0-4. 0 representing 'never experienced' and 4 representing 'almost always experienced'. Total score ranges between 0-20 with 0 representing never experiencing fatigue and 20 representing almost always experiencing fatigue.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 10.1 (1.22) | 8.7 (1.56)

22. Primary Outcome: Participant Fatigue Score - 5 Item Modified Fatigue Impact Scale.
Description: as for outcome 21
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Units on a scale | 6.6 (0.92) | 7.4 (1.83)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including both time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including both time points in the analysis

23. Secondary Outcome: Participant Muscle Tone Measure
Description: Myometer measured muscle tone taken from Erector Spinae muscle central belly via accelerometer probe registering response from a series of low force mechanical impulses applied perpendicular to the muscle. The muscle central belly was palpated while asking the participant to lift their head and feet at the same time while lying in prone position contracting this muscle. Measurements taken from a myometer device given as a frequency measure in Hertz. Further method details are given in the Protocol Document in attachments.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Hertz | 15.87 (1.48) | 13.2 (0.59)

24. Secondary Outcome: Participant Muscle Tone Measure
Description: as for outcome 23
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Hertz | 14.93 (0.84) | 13 (0.84)

25. Secondary Outcome: Participant Muscle Tone Measure
Description: as for outcome 23
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Hertz | 14.7 (1.05) | 12.83 (0.92)

26. Secondary Outcome: Participant Muscle Tone Measure
Description: as for outcome 23
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Hertz | 15.46 (1.17) | 12.78 (0.83)

27. Secondary Outcome: Participant Muscle Tone Measure
Description: as for outcome 23
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Hertz
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Hertz | 14.86 (1.1) | 12.32 (0.5)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Muscle tone values were analysed as a percentage change from baseline measurements to normalise group variances; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Muscle tone values were analysed as a percentage change from baseline measurements to normalise group variances; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

28. Secondary Outcome: Participant Muscle Elasticity Measure
Description: Myometer measured muscle elasticity taken from Erector Spinae muscle central belly via accelerometer probe registering response from a series of low force mechanical impulses applied perpendicular to the muscle. The muscle central belly was palpated while asking the participant to lift their head and feet at the same time while lying in prone position contracting this muscle. Measurements taken from a myometer device given as the logarithmic decrement of tissue's natural dampening frequency oscillation characterising its elasticity (dissipation of mechanical energy). Further method details are given in the Protocol Document in attachments.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Natural log of acceleration peak ratio
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Natural log of acceleration peak ratio | 1.36 (0.13) | 1.35 (0.1)

29. Secondary Outcome: Participant Muscle Elasticity Measure
Description: as for outcome 28
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Natural log of acceleration peak ratio
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Natural log of acceleration peak ratio | 1.51 (0.12) | 1.37 (0.14)

30. Secondary Outcome: Participant Muscle Elasticity Measure
Description: as for outcome 28
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Natural log of acceleration peak ratio
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Natural log of acceleration peak ratio | 1.39 (0.12) | 1.36 (0.13)

31. Secondary Outcome: Participant Muscle Elasticity Measure
Description: as for outcome 28
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Natural log of acceleration peak ratio
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Natural log of acceleration peak ratio | 1.34 (0.12) | 1.36 (0.13)

32. Secondary Outcome: Participant Muscle Elasticity Measure
Description: as for outcome 28
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Natural log of acceleration peak ratio
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Natural log of acceleration peak ratio | 1.43 (0.12) | 1.36 (0.13)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

33. Secondary Outcome: Participant Single Leg Stance Body Sway Anterior-Posterior Path Length
Description: Force plate recording from single leg stance balance test automatically outputted by software using centre of pressure recording to track position body sway travelled in the Anterior-Posterior position. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 343 (43.38) | 439.46 (56.91)

34. Secondary Outcome: Participant Single Leg Stance Body Sway Anterior-Posterior Path Length
Description: as for outcome 33
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 295.49 (23.98) | 381.02 (57.68)

35. Secondary Outcome: Participant Single Leg Stance Body Sway Anterior-Posterior Path Length
Description: as for outcome 33
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 260.85 (28.08) | 376.86 (55.14)

36. Secondary Outcome: Participant Single Leg Stance Body Sway Anterior-Posterior Path Length
Description: as for outcome 33
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 272.43 (25.31) | 357.17 (36.47)

37. Secondary Outcome: Participant Single Leg Stance Body Sway Anterior-Posterior Path Length
Description: as for outcome 33
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 279.76 (42.15) | 323.6 (37.3)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

38. Secondary Outcome: Participant Single Leg Stance Body Sway Medial-Lateral Path Length
Description: Force plate recording from single leg stance balance test automatically outputted by software using centre of pressure recording to track position body sway travelled in the Medial-Lateral position. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 275.19 (41.87) | 351.67 (56.61)

39. Secondary Outcome: Participant Single Leg Stance Body Sway Medial-Lateral Path Length
Description: as for outcome 38
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 282.06 (54.48) | 286.16 (41.95)

40. Secondary Outcome: Participant Single Leg Stance Body Sway Medial-Lateral Path Length
Description: as for outcome 38
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 223.9 (43.11) | 291.16 (51.78)

41. Secondary Outcome: Participant Single Leg Stance Body Sway Medial-Lateral Path Length
Description: as for outcome 38
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 211.89 (35.94) | 275.46 (45.11)

42. Secondary Outcome: Participant Single Leg Stance Body Sway Medial-Lateral Path Length
Description: as for outcome 38
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Millimeters
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters | 205.69 (37.69) | 296.17 (47.77)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

43. Secondary Outcome: Participant Single Leg Stance Body Sway Velocity
Description: Force plate recording from single leg stance balance test automatically outputted by software using centre of pressure recording to track position total body sway velocity travelled. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 49.02 (5.67) | 61.5 (7.66)

44. Secondary Outcome: Participant Single Leg Stance Body Sway Velocity
Description: as for outcome 43
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 45.36 (5.07) | 51.96 (6.48)

45. Secondary Outcome: Participant Single Leg Stance Body Sway Velocity
Description: as for outcome 43
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 38.42 (5.17) | 53.83 (7.25)

46. Secondary Outcome: Participant Single Leg Stance Body Sway Velocity
Description: as for outcome 43
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 37 (3.66) | 50.54 (5.07)

47. Secondary Outcome: Participant Single Leg Stance Body Sway Velocity
Description: as for outcome 43
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Millimeters/second
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Millimeters/second | 38.57 (5.52) | 48.77 (5.81)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis

48. Secondary Outcome: Participant Sit-to-Stand Rising Index
Description: Force plate recording from sit-to-stand test automatically outputted by software using percentage of body weight applied to the force plate during the stance phase of movement. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Percentage of Body Weight
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Percentage of Body Weight | 53.57 (4.89) | 56.98 (2.82)

49. Secondary Outcome: Participant Sit-to-Stand Rising Index
Description: as for outcome 48
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Percentage of Body Weight
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Percentage of Body Weight | 59.31 (4.99) | 60.92 (3.28)

50. Secondary Outcome: Participant Sit-to-Stand Rising Index
Description: as for outcome 48
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Percentage of Body Weight
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Percentage of Body Weight | 57.23 (4.04) | 58.99 (2.78)

51. Secondary Outcome: Participant Sit-to-Stand Rising Index
Description: as for outcome 48
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Percentage of Body Weight
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Percentage of Body Weight | 57.22 (3.12) | 59.33 (3.46)

52. Secondary Outcome: Participant Sit-to-Stand Rising Index
Description: as for outcome 48
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Percentage of Body Weight
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Percentage of Body Weight | 59.06 (2.28) | 61.53 (1.8)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p > 0.05, ANOVA — A priori threshold for statistical significance is 0.05; Repeated measures ANOVA including all 5 time points in the analysis

53. Secondary Outcome: Participant Sit-to-Stand Weight Transfer
Description: Force plate recording from sit-to-stand test automatically outputted by software using the time taken to reach full standing recorded by the force plate. Further details are outlined in the attached Protocol Document.
Time Frame: Taken at baseline, pre-treatment.
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Seconds | 3.83 (0.77) | 2.37 (0.13)

54. Secondary Outcome: Participant Sit-to-Stand Weight Transfer
Description: as for outcome 53
Time Frame: Taken immediately post 1st treatment, same day as baseline measures (week 1).
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Seconds | 2.4 (0.33) | 2.08 (0.13)

55. Secondary Outcome: Participant Sit-to-Stand Weight Transfer
Description: as for outcome 53
Time Frame: Taken immediately post 2nd treatment, 1 week after baseline measurements (week 2).
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Seconds | 2.83 (0.36) | 2.11 (0.23)

56. Secondary Outcome: Participant Sit-to-Stand Weight Transfer
Description: as for outcome 53
Time Frame: Taken immediately post 3rd treatment, 2 weeks after baseline measurements (week 3).
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Seconds | 2.69 (0.32) | 2.62 (0.2)

57. Secondary Outcome: Participant Sit-to-Stand Weight Transfer
Description: as for outcome 53
Time Frame: Taken immediately post 4th treatment, 3 weeks after baseline measurements (week 4).
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
Number analyzed (Participants) | 10 | 10
Seconds | 2.44 (0.21) | 2 (0.15)
Statistical Analysis 1: Comparison: Experimental A - Mobilisation Intervention; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis
Statistical Analysis 2: Comparison: Experimental B - General Massage; Test type: Superiority; p < 0.05, ANOVA — Including partial eta squared large effect size; Repeated measures ANOVA including all 5 time points in the analysis

ADVERSE EVENTS:
Time Frame: 4 testing sessions lasting 2 hours each, one week apart each time, lasting a total of 8 hours within a 3 week period.
Arm/Group | Experimental A - Mobilisation Intervention | Experimental B - General Massage
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Study was not able to recruit full number of participants required in the sample size calculation and large degree of variability exists within the population.

A longer term study with more treatment sessions may show more cumulative effect within the data results.

The study used an alternative treatment for group comparison rather than placebo for ethical and feasibility reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT05090709/Prot_SAP_000.pdf